CLINICAL TRIAL: NCT06411236
Title: Functional Response Characteristics of Brain Under Swallowing Task Paradigm Based on Functional Near-infrared Spectroscopy
Brief Title: Functional Response Characteristics of Brain Under Swallowing Task Paradigm
Status: Not yet recruiting | Type: Observational
Sponsor: Ruyao Liu (Other)
Responsible Party: Sponsor-Investigator, Ruyao Liu, Principal Investigator, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Other Study IDs: 2020-PT310-04
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Swallowing Disorder; Dysphagia; Swallowing Substances
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- middle and old group: A total of 15 middle-aged and elderly subjects were selected. Resting state detection: After entering the NIR assessment room, the subjects sat comfortably for 5 minutes, and then wore fNIRS headcaps. The subjects were asked to sit quietly and avoid moving and thinking for 30 seconds.
  Task state detection: Subjects entered the NIR assessment room, sat comfortably for 5 minutes, and then wore fNIRS headcaps. After resting for 30 seconds, the subjects were asked to swallow, swallow saliva for 20 seconds, rest for 20 seconds, and repeat three times.
- young group: A total of 15 young subjects were selected. Resting state detection: After entering the NIR assessment room, the subjects sat comfortably for 5 minutes, and then wore fNIRS headcaps. The subjects were asked to sit quietly and avoid moving and thinking for 30 seconds.
  Task state detection: Subjects entered the NIR assessment room, sat comfortably for 5 minutes, and then wore fNIRS headcaps. After resting for 30 seconds, the subjects were asked to swallow, swallow saliva for 20 seconds, rest for 20 seconds, and repeat three times.

SUMMARY:
Functional near-infrared spectroscopy was used to investigate the cortical activation patterns and lateralization during swallowing tasks in 15 healthy middle-aged and elderly people and 15 healthy young people. It provides a theoretical basis for the study of swallowing function and a new idea for the treatment of patients with swallowing disorders.

DETAILED DESCRIPTION:
Swallowing is coordinated by hyoid muscle group, pharyngeal muscle and upper esophageal muscle, as well as the regulation of swallowing related functional brain area. Dysphagia refers to the inability to safely and effectively transport food from the mouth to the stomach to obtain adequate nutrition and water, resulting in eating difficulties. Studies have shown that swallowing disorders are mainly caused by stroke, brain trauma, neurodegenerative diseases (Alzheimer's disease, Parkinson's disease, multiple sclerosis and amyotrophic lateral sclerosis) and head and neck cancers (oral tumors, nasopharyngeal and laryngeal cancers). Moreover, the prevalence of dysphagia increases with age. Patients with dysphagia often have many complications, which may lead to dehydration, malnutrition, aspiration, pneumonia, etc., which greatly delays the recovery process of patients and reduces the quality of life of patients. Studies have shown that the swallowing network includes multiple brain regions, including the primary somatosensory cortex, primary motor cortex, bilateral premotor and auxiliary motor cortex, cingulate cortex, prefrontal, temporal, precuneus, subparietal lobule, cerebellum and cerebellum.

At present, there are some functional near-infrared spectroscopy studies on the swallowing function of healthy people, which mainly focus on healthy young subjects, and studies show that the incidence of swallowing disorders increases with age, the incidence of swallowing disorders in people over 50 years old is 5.5% ~ 8%, and swallowing disorders are mainly concentrated in middle-aged and elderly people. At present, there are no studies on swallowing function in middle-aged and elderly healthy subjects with functional near-infrared spectroscopy. The purpose of this study is to explore and compare the cortical activation patterns and lateralization in the swallowing task of healthy middle-aged and elderly people and young people by using functional near-infrared spectroscopy, providing a theoretical basis for the exploration of swallowing function and further providing new ideas for the treatment of patients with swallowing disorders.

ELIGIBILITY:
Inclusion Criteria:

Middle and old age group: 50~70 years old; Young group: 18~25 years old; Right-handed; No history of neurological, psychiatric, respiratory, or swallowing dysfunction; No brain injury, epilepsy, head and neck disease, gastroesophageal reflux disease; No cases of skull defect, head infection and skin damage that could not be detected by function near-infrared spectroscopy; Subjects signed informed consent forms in accordance with the Declaration of Helsinki.

-

Exclusion Criteria:

pregnancy; poor patient compliance and non-cooperation with evaluation.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People aged 18-25 who met the inclusion exclusion criteria were included in the younger group. People aged 50-70 who met the exclusion criteria were included in the Middle aged group.Subjects need to understand the swallowing task and cooperate well.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-05-10 (Estimated); Primary Completion 2024-11-10 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
Functional near-infrared spectroscopy | day 1
  Resting state detection: After entering the NIR assessment room, the subjects sat comfortably for 5 minutes, and then wore fNIRS headcaps. The subjects were asked to sit quietly and avoid moving and thinking for 30 seconds.
  Task state detection: Subjects entered the NIR assessment room, sat comfortably for 5 minutes, and then wore fNIRS headcaps. After resting for 30 seconds, the subjects were asked to swallow, swallow saliva for 20 seconds, rest for 20 seconds, and repeat three times.

CONTACTS AND LOCATIONS:
Overall Officials: Xi Zeng, Study Chair — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The first affiliated hospital of zhengzhou university, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No
The datasets generated and analyzed during the current study are not publicly available due to the hospital's confidentiality regulations regarding trial data but are available from the corresponding author on reasonable request.